CLINICAL TRIAL: NCT07117344
Title: "Progranulin in Ankylosing Spondylitis Patients: A Potential Biomarker?"
Brief Title: Biomarkers in Ankylosing Spondylitis
Status: Recruiting | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Collaborators: Bilimsel Araştirma Projeleri Birimi, Istanbul Üniversitesi (Unknown)
Responsible Party: Principal Investigator, Seyda Sultan Eraslan, MD, Kirsehir Ahi Evran Universitesi
Other Study IDs: AhiEvranU-FTR-ŞSE-01
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Ankylosing Spondylitis (AS) / Radiographic Axial SpA (r-axSpA)
Keywords: ankylosing spondylitis; tnf; Progranulin; disease activity
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Blood samples taken from the patient will be centrifuged and stored as serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with ankylosing spondylitis on TNF inhibitors: Participants will be seen at one time and serum PGRN and TNF levels will be measured from each of them by ELISA method.
- patients with ankylosing spondylitis taking non-steroidal anti-inflammatory drugs: Participants will be seen at one time and serum PGRN and TNF levels will be measured from each of them by ELISA method.
- Control: Participants will be seen at one time and serum PGRN and TNF levels will be measured from each of them by ELISA method.

SUMMARY:
In this study, we aimed to compare serum PGRN(progranulin) and TNF-α levels in AS patients with healthy controls and to determine the relationship between TNF-α inhibitor use and PGRN levels in AS patients.

DETAILED DESCRIPTION:
Axial Spondyloarthritis is a heterogeneous group of diseases characterised by inflammatory low back pain, sacroiliitis, asymmetric oligoarthritis, dactylitis, enthesitis and uveitis.

The fact that PGRN acts by binding to TNF-α receptors, the use of TNF-α inhibitors in current treatment in patients with AS and the importance of this pathway in disease pathogenesis suggested that PGRN may be a marker associated with disease activity in these patients. In this study, we aimed to compare serum PGRN and TNF-α levels in patients with AS with healthy control group and to determine the relationship between TNF-α inhibitor use and PGRN levels in patients with AS.

In our study, 80 patients aged 20-65 years who were diagnosed with AS according to ASAS 2009 criteria and followed up in our clinic will be included. Patients with pregnancy or lactation status, acute or chronic infection findings, malignancy, and the presence of concurrent secondary rheumatic diseases other than AS will be excluded. As a healthy control group, 80 people aged 20-65 years without pregnancy or lactation, acute or chronic infection, malignancy and rheumatic disease will be recruited. Age, gender, comorbidities, duration of the disease, and medications used by all patients will be recorded. In addition, BASDAI, BASFI, BASMI, ASQoL, ASDAS-CRP, ESR, CRP levels will be recorded to determine the severity of AS clinically in the patient group. Participants in the patient and control groups will be seen at one time and serum PGRN and TNF levels will be measured by ELISA method.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 20-65
* Signing the informed consent form
* Axial spondyloarthropathy diagnosis according to ASAS 2009 criteria

Exclusion Criteria:

* Pregnancy or lactation
* Having signs of acute or chronic infection
* Presence of malignancy
* Having concurrent secondary rheumatic disease other than Axial Spondyloarthropathy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * Between the ages of 20-65
  * Signing the informed consent form
  * Axial spondyloarthropathy diagnosis according to ASAS 2009 criteria
  Exclusion Criteria:
  * Pregnancy or lactation
  * Having signs of acute or chronic infection
  * Presence of malignancy
  * Having concurrent secondary rheumatic disease other than Axial Spondyloarthropathy
  The healthy control group
  Inclusion Criteria:
  * Between the ages of 20-65
  * Signing the informed consent form
  Exclusion Criteria:
  Exclusion Criteria:
  * Pregnancy or lactation
  * Having signs of acute or chronic infection
  * Presence of malignancy or rheumatic diseases.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
In this study, we aimed to compare serum PGRN and TNF-α levels in AS patients with healthy controls and to determine the relationship between TNF-α inhibitor use and PGRN levels in AS patients. | Patient will be seen only once
  In this study, we aimed to compare serum PGRN and TNF-α levels in AS patients with healthy controls and to determine the relationship between TNF-α inhibitor use and PGRN levels in AS patients.

SECONDARY OUTCOMES:
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Patient will be seen only once
  Bath Ankylosing Spondylitis Disease Activity Index (BASDAI); BASDAI score consists of 6 questions. Patients are asked to give a score between 0 and 10 to each question as 'none' 0 points, 'very severe' 10 points according to their symptoms 1 week ago. Afterwards, the scores of the 5th and 6th questions are summed among themselves, divided by 2, added to the other scores and divided by 5 in total to obtain the BASDAI score. A BASDAI score of 4 and above indicates that the disease is out of control and that the patient's treatment, especially biological agents, should be reviewed. In the evaluation of response to treatment, a 50% improvement in the BASDAI score or a regression of at least 2 units on a 10-point scale is required
  Translated with DeepL.com (free version)
Ankylosing Spondylitis Disease Activity Scoring-CRP (ASDAS-CRP) | Patient will be seen only once
  Ankylosing Spondylitis Disease Activity Scoring-CRP (ASDAS-CRP) is a combined scoring system that measures disease activity. It is calculated by adding CRP value to clinical findings. According to the score obtained, disease activity is grouped as inactive, low, high and very high. In order to be considered for initiation of biological treatment, the ASDAS score must be at least 2.1. A change of 1.1 and above in the ASDAS score is considered a significant improvement, while changes of 2.0 and above are considered major improvements. For exacerbation in disease activity, there should be a change of 0.9 and above in the ASDAS score
Bath Ankylosing Spondylitis Functional Index (BASFI) | Patient will be seen only once
  Bath Ankylosing Spondylitis Functional Index (BASFI); patients are asked a total of 10 questions, including functional questions, and asked to score each question between 0 and 10, with 'easy' being 0 points and 'impossible' being 10 points. The score given to each question is summed and divided by 10 and the BASFI score is obtained .
Bath Ankylosing Spondylitis Metrology Index (BASMI) | Patient will be seen only once
  Bath Ankylosing Spondylitis Metrology Index (BASMI); metrological evaluation of patients is performed with this scoring. The score is calculated by measuring lumbar lateral flexion, tragus wall distance, modified schober test, cervical rotation and intermalleolar distance. It is used as a follow-up parameter in spinal mobility measurements
Ankylosing Spondylitis Quality of Life Scale (ASQoL) | Patient will be seen only once
  Ankylosing Spondylitis Quality of Life Scale (ASQoL) consists of 18 questions with a yes answer of 1 point and a no answer of 0 point. The score is calculated by summing the scores given to all questions. An increase in the score indicates poor quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No